CLINICAL TRIAL: NCT03775057
Title: Use of the MyDose Coach Digital Tool for Self-titration of Insulin in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Collaborators: Hospital Clinica Nova (Other)
Responsible Party: Principal Investigator, Dr. med. Hector Eloy Tamez Perez, Principal Investigator, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIE01-18
Record Dates: First submitted 2018-09-25; First posted 2018-12-13 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MyDose Coach app intervention (Experimental): The intervention involves the use of the MyDose Coach application, which has been previously programmed with the following titration scheme according to fasting glucose.
  Interventions: Other: MyDoseCoach app

INTERVENTIONS:
Other: MyDoseCoach app — The intervention involves the use of the MyDose Coach application, which has been previously programmed with the following titration scheme according to fasting glucose.

SUMMARY:
Scientific studies show that the introduction of digital tools led to: Significant improvement in glycemic control, greater patient satisfaction, reduction of emotional burden, reduction of fear of hypoglycaemia, reduction of anxiety of the regimen, significantly fewer of additional visits to the doctor in addition to those scheduled and a reduction of resources.

Primary Objective:

To evaluate the efficacy and safety of the MyDose Coach digital tool in patients with T2D with basal insulin or candidates for the use of basal insulin.

Secondary Objectives:

Evaluate demographic variables and control variables (HbA1c, SMPG, FPG). Measure the units of insulin used before and after the intervention

DETAILED DESCRIPTION:
The maximum study duration will be 29 weeks per patient that will consist of a 12-week screening period, a 16-week treatment period, and 1-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Greater than 18 years and up to 75 years of age
* Use of basal insulin once a day or candidate for basal insulin once a day based on% HbA1c according to international guidelines and doctor's criteria
* HbA1c > 7% in patients aged 18 to 65 years
* HbA1c > 7.5% in patients older than 65 years
* Patients who use basal insulin twice a day or premix with diagnosed hypoglycemia and who are candidates for switching from therapy to a basal insulin of one application per day
* Have a Smartphone
* Informed consent signature

Exclusion Criteria:

* Refuse to participate in the study.
* Age younger than 18 years old and over 75 years old.
* Diabetes type 1 or gestational (other than type 2 diabetes mellitus).
* Patients with the following chronic complications of diabetes: retinopathy and chronic kidney disease with a glomerular filtration rate <30 ml / min.
* The MyDose Coach tool is not appropriate for the patient or the use of the application is contraindicated (in the opinion of the Researcher, for example, patients with terminal illness, patients with cognitive or neurological disorders that are detailed below, patients who live alone and they do not have support from the family, patients with carpal tunnel who are not recommended to use a mobile phone, patients with musculoskeletal injuries in their hands, etc.)
* Patients who use insulin during the meal (short-acting analogue, regular human insulin or insulin premix) for more than 10 days in the last 3 months before the screening visit.
* Patients with severe hypoglycemia in the last 90 days.
* Hospitalization in the last 30 days (whatever the reason for hospitalization) In the last 3 months prior to the screening period: history of myocardial infarction, unstable angina, acute coronary syndrome, revascularization procedure, cerebrovascular accident requiring hospitalization.
* Severe or uncontrolled congestive heart failure (functional classification III and IV of the New York Heart Association [NYHA]).
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for a week or more within 90 days prior to the time of the test.
* Unable to meet specific protocol requirements (for example, inability to perform blood glucose measurements, administer your own insulin dose, or consider it unlikely that you will administer the titration safely according to your physician's guidance).
* Patients with cognitive disorders, dementia or any neurological disorder that affects the patient's ability to participate in the study, including the inability to understand the requirements of the study or to provide complete information about the adverse symptoms.
* Pregnant or breast-feeding women or women who intend to become pregnant during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-06-22 (Estimated); Study Completion 2019-08-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients reaching fasting SMPG target without a severe hypoglycemic episode during the 16-week on-treatment period | 16 weeks
  Percentage of patients reaching fasting SMPG (Self-Measured Plasma Glucose) target range 90-130 mg/dL (5.0-7.2 mmol/L) at Week 16 (mean of the last 4 readings recorded over the last 2 weeks) without a severe hypoglycemic episode (defined as having low blood glucose levels that requires assistance from another person to treat) during the 16-week on-treatment period

SECONDARY OUTCOMES:
Mean HbA1c change from baseline | 16 weeks
  Mean Glycated hemoglobin A1c (in percentage) from baseline
Percentage of patients reaching HbA1c of <7.5% and <7% | 16 weeks
  Percentage of patients reaching Glycated hemoglobin A1c of <7.5% and <7%
Mean fasting SMPG glucose change from baseline | 16 weeks
  Mean fasting Self-Measured Plasma Glucose (mean of the last 4 readings recorded over the last 2 weeks, in mg/dl)
Time to reach the first fasting SMPG target | 16 weeks
  Time in weeks to reach the first fasting SMPG target range of 90-130 mg/dL (5.0-7.2 mmol/L)
Mean FPG glucose change from baseline | 16 weeks
  Mean fasting plasma glucose glucose change from baseline, in mg/dl
Percentage of patients with hypoglycemic events | 16 weeks
  Percentage of patients with hypoglycemic events (blood glucose less than 70 mg/dL)
Number of hypoglycemic events | 16 weeks
  Number of hypoglycemic events (blood glucose less than 70 mg/dL)
Percentage of patients with adverse events | 16 week
  Percentage of patients with adverse events (other than hypoglycemia)
Assessment of emotional well-being using WHO-5 well-being index | 16 week
  Assessment of emotional well-being using WHO-5 well-being index. The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Nova, San Nicolás de los Garza, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided